CLINICAL TRIAL: NCT07322029
Title: Effect of Intrathecal Morphine on Quality of Recovery After Laparoscopic Gynecological Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, RenChun Lai, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025-FXY-311
Record Dates: First submitted 2025-12-08; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Laparoscopic Gynecological Surgery
Keywords: laparoscopic gynecological surgery; QoR-15; Intrathecal morphine
MeSH Terms: interventions — 1,3-bis(4-amidinophenoxy)-2-(4-amidinophenoxymethyl)ethylpropane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrathecal morphine group (Experimental): Before anesthesia induction, patients in the intervention group received an intrathecal injection of morphine at the L3-4 or L4-5 or L5-S1 interspace. The intrathecal morphine dose was 2 μg/kg.
  Interventions: Procedure: Intrathecal morphine group; Procedure: TAPB
- Normal saline group (Active Comparator): Before anesthesia induction, patients in the control group received an intrathecal injection of an equal volume of preservative-free normal saline at the L3-4 or L4-5 or L5-S1 interspace.
  Interventions: Procedure: Intrathecal saline injection; Procedure: TAPB

INTERVENTIONS:
Procedure: Intrathecal morphine group — With the patient in the lateral position, the puncture site was identified under ultrasound guidance. After local anesthesia, a spinal needle was advanced into the subarachnoid space, and intrathecal morphine was injected following confirmation of free cerebrospinal fluid flow.
  Arms: Intrathecal morphine group
Procedure: TAPB — With the patient supine, a linear ultrasound probe was placed between the costal margin and iliac crest to identify the abdominal wall layers. Using an in-plane approach, a needle was advanced into the transversus abdominis plane, and after negative aspiration, liposomal bupivacaine was injected under direct ultrasound visualization. The block was performed bilaterally.
  Arms: Intrathecal morphine group
Procedure: Intrathecal saline injection — With the patient in the lateral position, the puncture site was identified under ultrasound guidance. After local anesthesia, a spinal needle was advanced into the subarachnoid space, and an equal volume of preservative-free normal saline was injected after confirming cerebrospinal fluid flow.
  Arms: Normal saline group
Procedure: TAPB — With the patient supine, a linear ultrasound probe was placed between the costal margin and iliac crest to identify the abdominal wall layers. Using an in-plane approach, a needle was advanced into the transversus abdominis plane, and after negative aspiration, liposomal bupivacaine was injected under direct ultrasound visualization. The block was performed bilaterally.
  Arms: Normal saline group

SUMMARY:
Minimally invasive gynecologic surgery has become the standard approach for the treatment of benign and malignant gynecologic diseases, offering the advantages of reduced surgical trauma and faster recovery. However, postoperative pain remains a major barrier to optimal recovery, with up to 40% of patients experiencing moderate to severe pain within the first 24 hours after laparoscopic procedures. Laparoscopic gynecologic surgery typically induces both somatic pain from abdominal wall incisions and visceral pain caused by peritoneal traction and pneumoperitoneum, making effective analgesia challenging. Transversus abdominis plane block (TAPB) is commonly used to control somatic incisional pain but provides limited relief of visceral pain, often resulting in increased opioid consumption and opioid-related adverse effects such as dizziness and postoperative nausea and vomiting. Intrathecal morphine (ITM) offers potent and long-lasting visceral analgesia with minimal systemic opioid requirements and has demonstrated safety and efficacy across multiple surgical settings. The complementary analgesic mechanisms of TAPB and intrathecal morphine suggest that their combination may enhance postoperative recovery by improving pain control while reducing opioid use.

The objective of this randomized controlled trial is to evaluate whether the combination of intrathecal morphine and TAPB improves the quality of recovery after laparoscopic gynecologic surgery compared with TAPB alone. This study aims to provide high-quality clinical evidence to guide the development of an optimized multimodal analgesia strategy for patients undergoing minimally invasive gynecologic procedures.

DETAILED DESCRIPTION:
All patients will receive standardized general anesthesia combined with bilateral transversus abdominis plane block. The intervention group will additionally receive intrathecal morphine, whereas the control group will receive intrathecal saline. After entering the operating room, routine monitoring will include electrocardiography, pulse oximetry, noninvasive blood pressure, heart rate, and end-tidal carbon dioxide. Prior to anesthesia induction, patients in the intervention group will undergo lumbar intrathecal injection of morphine at the L3/4 or L4/5 or L5/S1 interspace. Based on previous literature and clinical experience, intrathecal morphine will be administered at a dose of 2 ug/kg. The control group will receive an equivalent volume of intrathecal normal saline under identical conditions.

General anesthesia will be induced with intravenous dexmedetomidine (0.5 ug/kg), Propofol (1.5-2 mg/kg), remifentanil (TCI 4 ng/mL), and rocuronium (0.6 mg/kg), followed by endotracheal intubation. Bilateral TAPB will be performed in all patients under ultrasound guidance. A total of 60 mL of diluted bupivacaine liposome (20 mL: 266 mg diluted to 60 mL with normal saline) will be administered, with 15 mL injected at each of the bilateral subcostal and lateral approaches (total 60 mL). Anesthesia maintenance will include 1.0-1.3 MAC desflurane, remifentanil, sufentanil, rocuronium, and vasoactive medications as required. Intraoperative opioid consumption will be recorded.

Postoperative analgesia will be provided using intravenous patient-controlled analgesia (PCA), consisting of 100 mg morphine diluted to a total volume of 100 mL. The PCA settings will include no background dose, a 1-mL bolus dose, and a 6-minute lockout interval. In cases of adverse events such as hypotension, fluid resuscitation and vasoactive support will be provided, and PCA parameters may be reduced or discontinued by an independent nurse if necessary.

The primary outcome of this study is the Quality of Recovery-15 (QoR-15) score at 24 hours postoperatively. Secondary outcomes include postoperative pain scores, opioid consumption, postoperative nausea and vomiting, pruritus, and other opioid-related adverse events. This trial aims to evaluate whether the combination of intrathecal morphine and TAPB provides superior analgesia and improves recovery after gynecologic laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged ≥18 years.
* Scheduled for elective laparoscopic gynecological surgery under general anesthesia.
* American Society of Anesthesiologists (ASA) physical status I-III.
* Able to provide written informed consent.

Exclusion Criteria:

* Contraindications to neuraxial anesthesia.
* Allergy to morphine or local anesthetics.
* Long-term opioid use (>20 morphine milligram equivalents per day).
* Baseline NRS pain score >3.
* Cognitive impairment or inability to cooperate.
* Emergency or non-elective surgery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligible participants must self-identify as female, as the surgical procedures under investigation apply only to female anatomy.
Enrollment: 252 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
QoR-15 score at 24 hours after surgery | 24 hours after surgery
  The Quality of Recovery-15 questionnaire is a validated patient-reported outcome measure assessing postoperative recovery across five domains (pain, physical comfort, emotional state, physical independence, and psychological support). Total scores range from 0 to 150, with higher scores indicating better quality of recovery.

SECONDARY OUTCOMES:
QoR-15 score at 48 and 72 hours postoperatively | 48 and 72 hours after surgery
  The QoR-15 total score ranges from 0 to 150, with higher scores indicating better quality of recovery.
Numeric Rating Scale (NRS) pain score at rest and cough at 24, 48, and 72 hours postoperatively | 24, 48, and 72 hours after surgery
  Pain intensity will be assessed using the Numeric Rating Scale, ranging from 0 (no pain) to 10 (worst imaginable pain), with higher scores indicating greater pain intensity.
Rest and cough NRS scores in post-anesthesia care unit (PACU) after surgery | 30 minutes after surgery
  Pain intensity will be assessed using the NRS, ranging from 0 to 10, with higher scores indicating greater pain intensity
Cumulative morphine equivalent consumption at 24, 48, and 72 hours postoperatively | 24, 48, and 72 hours after surgery
Time to first postoperative flatus | Up to 1 week after surgery
Time to first ambulation after surgery | Up to 1 week after surgery
  Time from surgery to the first postoperative ambulation.
Urinary catheter indwelling time | Up to 1 week after surgery
  Time from surgery to urinary catheter removal.
Time to first analgesic request | Up to 72 hours after surgery
Total amount of additional analgesic medication at 24, 48, 72 hours postoperatively | 24, 48, and 72 hours after surgery
Patient satisfaction assessed by a 0-100 numeric scale | At 72 hours after surgery
  Patient satisfaction with postoperative analgesia will be assessed using a numeric rating scale ranging from 0 to 100, where 0 indicates the lowest level of satisfaction and 100 indicates the highest level of satisfaction.
Length of hospital stay (days) | From surgery to hospital discharge
  Length of hospital stay is defined as the number of days from surgery to hospital discharge.
Incidence of postoperative shoulder pain assessed by the NRS | Up to 72 hours after surgery
  Postoperative shoulder pain will be assessed by patient report, defined as the presence of shoulder pain with a NRS score ≥1 during the postoperative period.
Incidence of adverse events at 24, 48, and 72 hours postoperatively | 24, 48, and 72 hours after surgery
  Postoperative adverse events include hypotension, dizziness, pruritus, and postoperative nausea and vomiting, assessed by clinical observation and medical records.
Incidence of chronic pain at 3 months and 6 months after surgery | 3 months and 6 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangdong, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No